CLINICAL TRIAL: NCT05264766
Title: The Use of Cooling Helmet for Neuroprotection Management in Patient Undergoing Open Heart Surgery: an Evaluation of Postoperative Neuron-specific Enolase (NSE) and Delirium
Brief Title: The Use of Cooling Helmet for Neuroprotection Management in Open Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Mohamad Prakoso Adji, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IndonesiaUAnes333
Record Dates: First submitted 2022-02-18; First posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Heart; Surgery, Heart, Functional Disturbance as Result
Keywords: cooling helmet; neuron specific enolase; delirium; open heart surgery
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cooling helmet on (Experimental): Cooling helmet on means there was circulating cold water inside the helmet, put after induction during cardiopulmonary bypass on
  Interventions: Device: Cooling helmet on
- Cooling helmet off (Active Comparator): Cooling helmet on means there was no circulating cold water inside the helmet, put after induction during cardiopulmonary bypass on
  Interventions: Device: Cooling helmet off

INTERVENTIONS:
Device: Cooling helmet on — Cooling helmet with circulating cold water
  Arms: Cooling helmet on
Device: Cooling helmet off — Cooling helmet without circulating cold water
  Arms: Cooling helmet off

SUMMARY:
To know the relationship between the use of cooling helmet with the changes of NSE level and postoperative delirium event in open heart surgery

DETAILED DESCRIPTION:
Subjects were assigned into two groups after giving consent to participate in the study using random allocation, 13 subjects per group. Blood sample from CVC were obtained to assess NSE preoperative. After induction, cooling helmet with circulating cold water were placed on patients group A and without circulating cold water on group B. Blood samples were obtain again 6 hours after cardiopulmonary bypass off to assess NSE postoperative. Delirium was assessed using Confusion Assessment Method - Intensive Care Unit (CAM-ICU)

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing their first open heart surgery using cardiopulmonary bypass
* Age ≥18 year-old
* Patient with American Society of Anesthesiologists (ASA) III
* Patient with Glasgow Coma Scale (GCS) 15, fully aware and oriented
* Patient fluent in Indonesia

Exclusion Criteria:

* Patients did not give consent to participate in the study
* Patients with central nervous system disease (stroke, intracranial tumor)
* Patients with psychiatric problem (schizophrenia, depression)
* Patients with cognitive problem
* Blind and deaf patient
* Patient on psychotrophic or narcotics medication

Drop out criteria

* Surgery without cardiopulmonary bypass
* Patient demise after surgery
* Patients decided to refrain from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Neuron-specific enolase | 6 hours post cardiopulmonary bypass off
  Neuronal injury marker. The higher the value, the worse the outcome
Confusion Assessment Method - Intensive Care Unit (CAM-ICU) | Changes of CAM-ICU from 12 hours to 24 hours postoperative
  Tools to assess delirium. The higher the errors, the worse the outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Central National Hospital, Jakarta Pusat, DKI Jakarta, Indonesia